CLINICAL TRIAL: NCT04474756
Title: Comparison of Efficacy of Two Mandibular Advancement Devices (MADs) and Insights Gain From Analysis of Mandibular Behavior During Sleep
Brief Title: Comparison of Efficacy of Two Mandibular Advancement Devices (MADs) During Sleep
Acronym: SONAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A01714-53
Record Dates: First submitted 2019-12-26; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Apnea Syndrome
Keywords: Obstructive Sleep Apnea; mandibular advancement devices; Mandibular movement; Polysomnography
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, comparative, open, multicenter study. 90 patients, randomized into two parallel groups, comparing the efficacy of 2 different custom-made mandibular advancement devices: NarvalTM versus TALITM, in the treatment of obstructive sleep apnea (OSA).
Masking Description: open, multicenter study in 90 obstructive sleep apnea (OSA) patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandibular Advancement Devices Narval™ (Experimental): The tested device Narval™ will be a custom-made adjustable bi-block mandibular advancement device, that is made with semi-rigid plastic materials (bio-compatible polymer) and customized using a high-precision computer-aided design (CAD)/computer-aided manufacturing (CAM) ) (ResMed, Narval CC™). The Mandibular Advancement Devices will be gradually adjusted to provide mandibular advancement over a 15-mm range. Each Mandibular Advancement Device will be ﬁtted by a dental specialist with an initial advancement of about 60 % of maximal jaw protrusion. During titration, mandibular advancement will be adjusted at the discretion of the dental specialist.
  Interventions: Device: custom-made adjustable mandibular advancement device
- Mandibular Advancement Devices TALI ™ (Active Comparator): The control device TALI ™ is a mandibular advancement orthesis, customized and manufactured by the "laboratoire TALI", of the bi-bloc type consisting of rigid gutters thermo-formed on the plaster dental arches and articulated by two links of variable size allowing to adjust the advance in steps of 1 millimeter. This orthesis is manufactured on molding from bio-compatible plastic materials. The different sizes of rods proposed allow mandibular advances of 4 mm to 16 mm. Two clinical studies evaluated the effectiveness of the AMC / AMO orthosis (initial version of the TALI orthesis, with non-curved links) in patients with OSA. They have already demonstrated the effectiveness of the TALI orthesis by decreasing AHI and drowsiness; most patients preferred to use the orthesis (76.4% vs. 9.1%)11.
  Interventions: Device: custom-made adjustable mandibular advancement device

INTERVENTIONS:
Device: custom-made adjustable mandibular advancement device — a custom-made mandibular repositioning device (MRD), available under medical prescription for the treatment of adult obstructive sleep apnea (OSA) and snoring. It maintains the mandible in an advanced position along the occlusal plane. This ensures patient comfort and treatment efficacy.
  Other Names: mandibular advancement orthosis (MAD)

SUMMARY:
Mandibular Advancement Devices (MADs) are now a reliable alternative to continuous positive airway pressure (CPAP) treatments for Obstructive Sleep Apnea (OSA) . Despite good tolerance and efficacy, there are still barriers limiting the widespread use of MAD and its acceptance in OSA routine clinical practice. Various MAD designs currently exist and constantly emerge on the market without clear evidence regarding the best technical choice and the cost-effectiveness compromise. Although these MAD has been tested in term of efficacy, no study has tested the difference between MADs in term of efficacy, tolerance and patient satisfaction. The aim of this clinical trial is to compare the effectiveness of two MADs - custom-made titratable MAD (NarvalTM) and customizable titratable MAD (TALITM), over a 3-month period, in patients with obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is characterized by repetitive episodes of partial or complete pharyngeal obstruction during sleep. OSA is one of the most frequent chronic diseases with both social and multi-organ consequences making it an economic burden for society. OSA durably impairs the quality of life of patients and their entourage and is associated with co-morbidities including hypertension, arrhythmias, stroke, coronary heart disease and metabolic dysfunction.

Continuous positive airway pressure (CPAP), the first line therapy for OSA, requires high adherence to be effective in terms of symptom improvement and reduction of the burden of co-morbidities. For one third of patients, such adherence is difficult to achieve in the long term and mandibular advancement devices (MAD) have emerged as the leading alternative to CPAP. So, MADs are now a reliable alternative to CPAP treatments, which position these in numerous patients as a first therapy. Moreover, mild to moderate symptomatic patients who refuse to be diagnosed are now referring to sleep centers in order to be treated. MAD and CPAP are similarly effective on symptoms, quality of life and in attaining reductions in blood pressure and cardiovascular morbidity. Although CPAP has a greater effect on Apnea + hypopnea index (AHI) reduction, adherence is better with MAD explaining the comparable mean disease alleviation achieved by the two treatment modalities.

Despite good tolerance and efficacy, there are still barriers limiting the widespread use of MAD and its acceptance in OSA routine clinical practice. Various different MAD designs currently exist and constantly emerge on the market without clear evidence regarding the best technical choice and the cost-effectiveness compromise. Titratable two-piece custom-made MADs are the gold standard in clinical guidelines and several brands are now on the market. Although these MAD has been tested in term of efficacy, no study has tested the difference between MADs in term of efficacy, tolerance and patient satisfaction. Such a paradigm merits being tested in a randomized controlled trial. The SONAR study is a multicenter, parallel-group randomized controlled trial to determine if the titratable MAD NARVAL TM is superior to the titratable MAD TALITM in OSA patients eligible for MAD. The primary outcome will be the treatment response at 3 months assessed by the difference of delta AHI at baseline and follow-up measured by polysomnography and secondary outcomes focus at global efficacy, tolerance and patient satisfaction.

To our knowledge it will be the first study comparing two titrable MADs.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before participation
2. Age ≥18 years
3. Moderate to severe OSA defined by:

   * AHI ≥30 or,
   * 15≤ AHI <30, but associated with excessive daytime sleepiness or,
   * 15≤ AHI <30, with at least two of the following criteria not explained by other factors: severe and daily snoring, choking or suffocating sensation during sleep, non-restorative sleep, daytime fatigue, difficulty concentrating, nocturia (more than one urination per night).
4. Naïve from any mandibular advancement device
5. Patient affiliated to a social security/health insurance system

Exclusion Criteria:

1. One or more of the following contra-indications:

   * dental problems (tooth failure, poor distribution or insufficient dental retention)
   * periodontal problems: active periodontitis not stabilized. Presence of periodontal pockets, advanced bone loss, significant tooth mobility, insufficient dental plaque control.
   * temporomandibular joint disorder (TJD)
   * maximum mandibular propulsion distance limited (< 6 mm)
2. More than 20% of central apnea and hypopnea
3. Severe psychiatric or neuromuscular disorder
4. Body Mass Index (BMI) > 30 kg/m2
5. Current orthodontic treatment or planned during the study
6. Pregnant women based on clinical exam and medical questioning.
7. Subject in exclusion period of another interventional study
8. Subject under administrative or judicial control
9. Subject unable to understand, follow objectives or methods due to cognition or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of efficacy of two Mandibular Advancement Devices: NarvalTM and TALITM | at the end of the 3-month period
  The difference of effectiveness between Mandibular Advancement Devices will be assessed using the difference of delta AHI, measured by Polysomnography, between the visit 2 (M3) and the Polysomnography before Mandibular Advancement Devices installation.

SECONDARY OUTCOMES:
To compare the efficacy of titration with each Mandibular Advancement Devices | between the oral appliance delivery and the end of the titration period at 3 months
  Delay of titration period, number of additional titration visits required
To compare the number of patients appropriately treated by Mandibular Advancement Devices between the two devices | after 3 months of treatment with mandibular advancement device
  Rate of complete response (AHI<10) or partial response (AHI<15) of treatment:
  The percentage of patients with AHI <15, or ≥ 50% reduction in AHI from baseline (D0) to D90 (3 months), associated with a subjective (patient reported) compliance ≥ 5 nights/week and 5 hours/night. AHI assessed by polysomnography
To compare the tolerance in the 2 arms | after 3 months of treatment
  Rate of side effects, jaw discomfort (visual analogic scale) scale), mean number of hours by night wearing the mandibular device (patient diary), therapy withdrawals
To compare the sleep quality | after 3 months of treatment with mandibular advancement device
  RDI, total sleep time, TST, PST, Sleep latency, WASO, Sleep efficiency, Time in stage I, II, SWS and REM sleep respectively, Total micro-arousals, respiratory micro-arousals and PLM micro-arousals, assessed by Polysomnography.
To compare the mandible behavior (mandibular movement (MM)) during sleep) with each Mandibular Advancement Device | after 1 month and 3 month of treatment with each Mandibular Advancement Device
  Mandibular movement, RDI and time spent in respiratory effort, assessed by home-based recording (by Class IIA polygraphic device: Sunrise® Solution with mandibular movement recording), and mandibular movement recording by Jaw-ac technology, added to the classical procedure (Polysomnography)
To compare the evolution of obstructive sleep apnea associated subjective daytime sleepiness with each Mandibular Advancement Device | after 3 months of treatment with each Mandibular Advancement Device
  by Epworth sleepiness score
To compare subjective snoring perception by the patient's environment | after 3 months of treatment with each Mandibular Advancement Device
  by subjective snoring (visual analogic scale-VAS)
To compare patient satisfaction | after 3 months of treatment with mandibular advancement device
  using the Questionnaire VSQ-VF
To compare the effect of obstructive sleep apnea on patient's quality of life | after 3 months of treatment with each Mandibular Advancement Device
  by Quebec Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Renaud TAMISIER, MD, PhD, Principal Investigator — Grenoble University Hospital, La Tronche 38700, France,
Locations (1):
- Grenoble University Hospital, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: No